CLINICAL TRIAL: NCT04896788
Title: Monitoring of the Post-vaccination Immune Response to COVID-19 Among Hospital Staff
Acronym: COVIDIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RBHP 2021 HENQUELL
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Hospital Staff; Vaccined Againt COVID-19
Keywords: Humoral response to Covid-19 Vaccine; Cellular response to Covid-19 Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monitoring of the immune response (Other): Immune response controlled with blood sample at 3, 6, 12, 18 and 24 months
  Interventions: Biological: Monitoring of the immune response

INTERVENTIONS:
Biological: Monitoring of the immune response — Blood sample at 3,6,12,18 and 24 months in order to assess the blood level of anti-S1 / RBD anticoprs

SUMMARY:
Vaccination against COVID-19 is a major public health issue to control the epidemic and reduce the number of severe infections and deaths. Three vaccines currently received use authorization in France: two mRNA vaccines and one recombinant viral vector vaccine. Immunogenicity data demonstrate that they induce the development of neutralizing antibodies and IgG directed against the viral S1 protein and the receptor binding domain (RBD). However, there are currently no data on the persistence over time of the humoral response induced by vaccination, and data are still incomplete on cellular immunogenicity. No immune correlate of protection has been established for COVID-19.

In addition, these data come from assays carried out with current vaccines developed against a lineage of SARS-CoV-2 known as wild type (without genetic mutations).

The main objective of this study is to monitor in hospital staff the temporal evolution of humoral immunity induced by anti-COVID-19 vaccines by using enzyme-linked immunosorbent assays (ELISA), at 3, 6, 12 and 24 months after the last injection of vaccine.

DETAILED DESCRIPTION:
* All medical, para-medical, medico-technical and administrative staff of the Clermont-Ferrand university hospital will be informed of the protocol through intra-hospital communication. The inclusion visit will be scheduled within 3 months +/- 14 days after the last injection of the vaccine. For volunteers who have not received their first injection, they will be offered to participate in the sub-study including an additional visit on the day of vaccination. They will be free to accept or refuse.
* As recruitment is consecutive, an anonymous list of potentially eligible subjects (with demographic data: age, sex; nature of the vaccine received) will be kept, in order to verify afterwards if the sample is representative.
* The study includes:

  1. Five visits over 21 months, 6 over 24 months for the subgroup included on the day of vaccination
  2. An interview with an investigator during the first visit, to collect the following data: hospital function, age, sex, weight, height, possible comorbidities exposing to a serious COVID-19 infection, possible COVID-19 infection prior to vaccination, date of vaccination and type of vaccine
  3. A self-questionnaire to update clinical data if necessary during the following visits
  4. A blood test at each visit, i.e. 2 tubes of 5 mL (antibody assays) and 4 tubes of 1 mL (cellular immunity assay).

     Blood samples will be stored at -80°C, before destruction at the end of the study.
* In the case of suspecting symptoms of COVID-19 during follow-up, molecular testing of SARS-CoV-2 infection will be offered and performed from nasopharyngeal swab or saliva sample.

ELIGIBILITY:
Inclusion Criteria:

* Adult person, man or woman, staff of the Clermont-Ferrand University Hospital (medical or paramedical, medico-technical or administrative caregiver), having received the second dose of vaccine (or the single dose if the single-dose vaccination schedule) against COVID- 19 3 months +/- 15 days before the inclusion visit, as part of the national vaccination campaign, regardless of the type of vaccine administered.
* For the subgroup included before vaccination (study of the pre-vaccination cellular response): Adult person, man or woman, staff of Clermont-Ferrand University Hospital (medical or paramedical, medico-technical or administrative caregiver), receiving the 1st injection on the same day or in the 7 days before the inclusion visit, regardless of the type of vaccine administered
* Commitment to respect the schedule of visits provided for in the research protocol
* Able to give informed consent to participate in research
* Affiliation to a social security scheme

Exclusion Criteria:

* Pregnancy or breastfeeding in progress at inclusion, or planned during follow-up
* Person under guardianship, guardianship or legal protection
* Whether the vaccine received was experimental or not authorized
* Refusal of participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-05-19 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
the blood level of anti-S1 / RBD antibodies | 3 months
  temporal evolution of humoral immunity induced by the anti-COVID-19 vaccine, at 3, 6, 12 and 24 months after the second injection (or the single injection if single dose vaccination schedule), using two quantitative enzyme-linked immunosorbent assays (ELISA) targeting anti-S1 and anti-RBD antibodies.
the blood level of anti-S1 / RBD antibodies | 6 months
  temporal evolution of humoral immunity induced by the anti-COVID-19 vaccine, at 3, 6, 12 and 24 months after the second injection (or the single injection if single dose vaccination schedule), using two quantitative enzyme-linked immunosorbent assays (ELISA) targeting anti-S1 and anti-RBD antibodies.
the blood level of anti-S1 / RBD antibodies | 12 months
  temporal evolution of humoral immunity induced by the anti-COVID-19 vaccine, at 3, 6, 12 and 24 months after the second injection (or the single injection if single dose vaccination schedule), using two quantitative enzyme-linked immunosorbent assays (ELISA) targeting anti-S1 and anti-RBD antibodies.
the blood level of anti-S1 / RBD antibodies | 24 months
  temporal evolution of humoral immunity induced by the anti-COVID-19 vaccine, at 3, 6, 12 and 24 months after the second injection (or the single injection if single dose vaccination schedule), using two quantitative enzyme-linked immunosorbent assays (ELISA) targeting anti-S1 and anti-RBD antibodies.

SECONDARY OUTCOMES:
relationship between the level of antibodies detected by serological tests (ELISA) and the antibodies titrated using an in vitro neutralization test | 3 months, 6 months, 12 months, 18 months, 24 months
  Comparison of the humoral response evaluated by serological tests with that analysed by neutralisation in vitro, on pairs of samples chosen to cover the variability of the response induced by vaccination between M3 and M24.
anti-S lymphocyte response induced by the anti-COVID-19 vaccine | 3 months, 6 months, 12 months, 18 months, 24 months
  Cellular immune response induced by the anti-COVID-19 vaccine evaluated by the anti-S lymphocyte response reflected by the determination of IFN-γ at the 3rd, 6th, 12th, 18th and 24th months after the second injection of vaccine (or the single injection if scheme single dose vaccine).
effect of age on immune response | 3 months, 6 months, 12 months, 18 months, 24 months
  Study the effect of age on the various immune parameters studied, in general and in their temporal course
Intensity of immune response according to different comorbidities | 3 months, 6 months, 12 months, 18 months, 24 months
  Study the effect of comorbidities on the various immune parameters studied, in general and in their temporal course
Intensity of immune response according to a previous COVID-19 infection or not | 3 months, 6 months, 12 months, 18 months, 24 months
  Study the effect of a previous COVID-19 infection on the various immune parameters studied, in general and in their temporal course
Intensity of immune response according to the type of vaccine administered | 3 months, 6 months, 12 months, 18 months, 24 months
  Study the effect of the type of vaccine administered on the various immune parameters studied, in general and in their temporal course
the cellular immune response directed against the Spike peptides of T lymphocytes before vaccination, between D-7 and the day of the 1st injection of vaccine | Day 1
  Pre-vaccine anti-S cellular immune response reflected by the IFN-γ assay, for a subgroup of 50 volunteers then benefiting from the same follow-up until the 24th month
genomic characteristics of the strain of SARS-CoV-2 in case of proven COVID-19 infection during follow-up | up to 24 months
  Clinical description of subjects presenting with COVID-19 infection during follow-up, and genomic characteristics of their strain of SARS-CoV-2 by whole genome sequencing (next-generation sequencing).

CONTACTS AND LOCATIONS:
Locations (1):
- Clermont-Ferrand University Hospital, Clermont-Ferrand, AURA, France

REFERENCES:
- [Derived] Bonnet B, Chabrolles H, Archimbaud C, Brebion A, Cosme J, Dutheil F, Lambert C, Junda M, Mirand A, Ollier A, Pereira B, Regagnon C, Vidal M, Evrard B, Henquell C. Decline of Humoral and Cellular Immune Responses Against SARS-CoV-2 6 Months After Full BNT162b2 Vaccination in Hospital Healthcare Workers. Front Immunol. 2022 Mar 2;13:842912. doi: 10.3389/fimmu.2022.842912. eCollection 2022. PMID 35309363